CLINICAL TRIAL: NCT03730038
Title: Effects of Pitavastatin Treatments on the Plasma Lgi3 Level in the Patients With Dyslipidemia: A Randomized Crossover Trial
Brief Title: Effects of Pitavastatin Treatments on the Plasma Lgi3 Level in the Patients With Dyslipidemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 4-2018-0794
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Dyslipidemias
Keywords: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Intervention Model Description: Patients who assigned to the pitavastatin treatment first group will be given the pitavastatin, followed by wash-out period and life-style modification treatment. Patients who assigned to the life-style modification treatment first group, will be treated with life-style modification treatment first, followed by wash-out period and pitavastatin treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pitavastatin treatment (Experimental): Treatment of pitavastatin 4 mg qd for 12 weeks
  Interventions: Drug: Treatment of pitavastatin 4 mg qd for 12 weeks
- Life-style modification (Active Comparator)
  Interventions: Behavioral: Life-style modification

INTERVENTIONS:
Drug: Treatment of pitavastatin 4 mg qd for 12 weeks — Treatment of pitavastatin 4 mg qd for 12 weeks
  Arms: Pitavastatin treatment
Behavioral: Life-style modification — Nutritional support with the meal less than 65% of carbohydrate, less than 30% of fat. Exercise 3-4 times, 30 min
  Arms: Life-style modification

SUMMARY:
Leucine-rich glioma inactivated 3(Lgi3) has been postulated to have a pro-inflammatory adipokine that inter-plays with other adipokines in adipogenesis and metabolic inflammation according to recent investigations. Thus, in this study, we sought to demonstrate that the treatment of statin can decrease Lgi3 level along with the decrease of the atherosclerosis to further evaluate the role of Lgi3 in atherosclerosis.

DETAILED DESCRIPTION:
Patients who assigned to the pitavastatin treatment first group will be given the pitavastatin 4 mg qd treatment for 12 weeks after randomization, followed by wash-out period of 3 weeks and life-style modification treatment for 12 weeks. Similarly, patients who assigned to the life-style modification treatment first group, will be treated with life-style modification treatment for 12 weeks after randomization, followed by wash-out period of 3 weeks and pitavastatin treatment for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-80 years
* Patients with intermediate or low cardiovascular risks needing the statin treatment
* Patients with intermediate or low cardiovascular risks treating the statin treatment

Exclusion Criteria:

* Patients without signed informed consent
* Patients with myopathy
* Pregnant women or women with potential childbearing
* Patients with diabetes
* Patients with established coronary artery disease
* Patients with heart failure
* Life expectancy less than 1 year

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Changes in Lgi3 level | At 12 weeks after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided